CLINICAL TRIAL: NCT04588987
Title: A Study to Evaluate the Safety and Efficiency of Using the Neoadjuvant Therapy With Carilizumab and Apatinib in Patients With Recurrent High-Grade Glioma ：A Prospective, Randomized Study
Brief Title: Neoadjuvant Carilizumab and Apatinib for Recurrent High-Grade Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongping Chen, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GBM-II-001
Record Dates: First submitted 2020-09-06; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Neoadjuvant Therapy; Carilizumab; Apatinib; Recurrent High-Grade Glioma
MeSH Terms: conditions — Glioma | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant group (Experimental): Patients need to treat with PD-1 and apatinib before surgery. Sequential therapy with PD-1 and apatinib when patients accepted surgery.
  Interventions: Biological: PD-1
- Adjuvant group (Experimental): Before surgery, patients no need to treat with PD-1 and apatinib. Sequential therapy with PD-1 and apatinib when patients accepted surgery.
  Interventions: Biological: PD-1

INTERVENTIONS:
Biological: PD-1 — Neoadjuvant PD-1 and Apatinib for rHGG. Adjuvant PD-1 and Apatinib for rHGG
  Other Names: apatinib

SUMMARY:
GBM is the most common intracranial tumor in adults, accounting for about 40% of all primary intracranial tumors.Although surgery, radiotherapy and chemotherapy have been used, the prognosis of glioma patients is still very poor. The study aim to Evaluate the Safety and efficiency of Using the neoadjuvant therapy with Carilizumab and Apatinib in patients with Recurrent High-Grade Glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age 18-70 years old, both male and female.
3. After biopsy or surgery, the postoperative pathological diagnosis was WHO III-IV glioma.
4. Patients in whom surgery can be safely delayed for a minimum period of 2 weeks following the administration of the first dose of nivolumab, in the opinion of the investigator.
5. KPS score ≥60；
6. Life expectancy >12 weeks.
7. Adequate organ function defined by:

   1. HGB≥110g/L；
   2. WBC≥3.0×109/L；NEUT≥1.5×109/L；
   3. PLT ≥75×109/L；

   <!-- -->

   1. BIL≤1.5ULN；
   2. ALT and AST≤2.0×ULN；
   3. creatinine < 1.5 x ULN or estimated creatinine clearance≥50ml/min（using the Cockcroft-Gault formula）

Exclusion Criteria:

1. Presence of extracranial disease.
2. Previous treatment with a PD-1, PDL-1 or CTLA-4，VEGFR targeted therapy.
3. Pregnant or breastfeeding patients.
4. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Routine testing is not required.
5. Positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.
6. History of allergy to study drug components or of severe hypersensitivity reactions to any monoclonal antibodies.
7. Known drug or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 3 years
  Time from enrollment to the dates of death from any cause or last follow up reported between date of first patient enrollment

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 18 months
  Time from enrollment to the dates of disease progression,death from any cause or last tumor assessment reported between date of first patient enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer center of Sun Yat sen University, Guangzhou, Guangdong, China